CLINICAL TRIAL: NCT05767827
Title: Effect of Dexmedetomidine As Adjuvant to Ropivacaine for Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nepal Medical College and Teaching Hospital (Other)
Responsible Party: Principal Investigator, Rajiv Yadav, Lecturer, Nepal Medical College and Teaching Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NepalMCTH
Record Dates: First submitted 2023-02-14; First posted 2023-03-14 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Local Anesthesia Adjuvants; Upper Extremity Fracture; Brachial Plexus Block
MeSH Terms: interventions — Ropivacaine; Lidocaine; Epinephrine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group R (Active Comparator): 0.35% ropivacaine 20ml, 1.5% lidocaine with adrenaline 10ml = 30 ml
  Interventions: Drug: ropivacaine, lidocaine with adrenaline
- Group RD (Experimental): 0.35% ropivacaine and 1mcg/ kg dexmedetomidine (20 ml), 1.5% lidocaine with adrenaline (10ml) = 30 ml
  Interventions: Drug: Dexmedetomidine, ropivacaine, lidocaine with adrenaline

INTERVENTIONS:
Drug: ropivacaine, lidocaine with adrenaline — Group R includes 0.35% ropivacaine 20ml, 1.5 % lidocaine with adrenaline 10ml
  Arms: Group R
Drug: Dexmedetomidine, ropivacaine, lidocaine with adrenaline — Dexmedetomidine 1mcg/kg and 0.35% ropivacaine with normal saline (20ml), 1.5% lidocaine with adrenaline (10ml) in group RD
  Arms: Group RD

SUMMARY:
Brachial plexus block is used for upper limb surgery. Local anesthesia alone for brachial plexus block provides good operative conditions, but have short duration of postoperative analgesia. Hence, various adjuvants to local anaesthetic agents to prolong the duration of peripheral nerve, analgesia. However, results are either inconclusive or associated with side effects. The purpose of this study is to determine whether dexmedetomidine as an adjuvant to ropivacaine in brachial plexus block improve quality of block in terms of duration of post operative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and II patients, weight 45 to 74 kg
* Elective upper limb surgery under brachial plexus block

Exclusion Criteria:

* known hypersensitivity or contraindication to ropivacaine, lidocaine and dexmedetomidine
* Pregnant or lactating mothers
* Hepatic, renal or cardiopulmonary abnormalities
* Long term analgesic therapy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Assess the duration of analgesia after brachial plexus block with ropivacaine and dexmedetomidine | 5 months
  Analgesia will be assessed with the help of Visual analogue score ( VAS). VAS greater than 3 will be given inj.ketorolac 30mg IV.
Assess the onset of sensory and motor block after brachial plexus block with ropivacaine and dexmedetomidine | 5 months
  Sensory block assessed by 3point scale
  0 normal sensation
  1. loss of sensation of pinprick
  2. loss of sensation of touch Duration of sensory block, defined as time interval between complete sensory block and complete resolution of anesthesia (score 0).Motor blockade assessed by modified Bromage scale (MBS)
  0-able to raise extended arm to 90 degree for full two seconds
  1. able to flex elbow, move fingers but unable to raise extended arm
  2. unable to flex elbow but able to move fingers
  3. unable to move arm, elbow, fingers Duration of motor block defined as time interval from complete motor block to recovery of complete motor function (MBS 0).
Assess the duration of sensory and motor block after brachial plexus block with ropivacaine and dexmedetomidine | 5months
  Duration of sensory block, defined as time interval between complete sensory block and complete resolution of anesthesia (score 0).
  Duration of motor block defined as time interval from complete motor block to recovery of complete motor function (MBS 0).

SECONDARY OUTCOMES:
Assess any complications of study drugs | 5 months
  Complications like bradycardia assessed by continue ECG monitoring, Hypotension will be assessed by NIBP

CONTACTS AND LOCATIONS:
Locations (1):
- Nepal medical college, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No